CLINICAL TRIAL: NCT04878328
Title: Leveraging Community Health Workers to Improve COVID-19 Testing and Mitigation Among Criminal Justice-involved Individuals Accessing a Corrections-focused Community-based Organization
Brief Title: Leveraging CHWs to Improve COVID-19 Testing and Mitigation Among CJIs Accessing a Corrections-focused CBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: The Fortune Society (Unknown); University of Bristol (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Cepheid (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2021-12976; 5R01MD016744 (NIH)
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Covid19
Keywords: COVID19; justice-involved individuals; Point-of-care testing; community based organization
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a randomized trial to assess the effectiveness of an onsite Point-of-Care testing and education intervention (O-PoC) compared to standard of care (SoC) at The Fortune Society (Fortune). The current SoC includes a referral to offsite community testing. Guided by Social Cognitive Theory, in O-PoC we will employ CHWs with lived experience of incarceration to provide: 1) COVID-19 education; 2) SARS-CoV-2 testing with Cepheid XpertXpress PCR tests at Fortune facilities; 3) Needs assessments and facilitated access to masks and hygiene supplies; 4) Navigation to vaccination sites (when available) and single-room housing at Fortune's supportive housing sites and partnering shelters, or alternative strategies that will maximize the ability to socially distance for those who test PCR positive; 5) Supportive counseling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- onsite Point-of-care (o-POC) (Experimental): CHWs will reach out to participants to schedule O-PoC visits. At O-PoC visits, CHWs will provide: 1. COVID-19 education; 2. PoC Cepheid XpertXpressSARS-CoV-2PCR tests; 3. Needs assessments and facilitated access to masks and hygiene supplies; 4. Navigation to vaccination sites (when available) and single-room housing at Fortune's supportive housing sites and partnering shelters or alternative strategies that will maximize the ability to socially distance for those who test PCR positive; 5. Supportive counseling. Due to SCT's emphasis on social influence, external and internal social reinforcement, we propose our O-PoC intervention delivered by CHWs onsite at Fortune locations over a 12-month period will lead to increased uptake of mitigation behaviors.
  Interventions: Behavioral: Onsite Point-of-care
- Standard of Care (SOC) (No Intervention): The current standard of care (SoC) for SARS-CoV-2 testing for Fortune clients is referral to offsite community testing sites and informal, unstructured education. In the SoC arm, Fortune staff will provide clients with a list of offsite SARS-CoV-2 testing locations, which are published online and available to all NYC residents. Those without insurance are not subject to a copay. Participants in SoC will continue to receive Fortune's suite of services as they are delivered (remote and/or in-person) at the time of study participation.

INTERVENTIONS:
Behavioral: Onsite Point-of-care — Guided by Social Cognitive Theory, O-PoC will employ CHWs with lived experience of incarceration to provide: 1) COVID-19 education; 2) SARS-CoV-2 testing with Cepheid XpertXpress PCR tests at Fortune facilities; 3) Needs assessments and facilitated access to masks and hygiene supplies; 4) Navigation to vaccination sites (when available) and single-room housing at Fortune's supportive housing sites and partnering shelters, or alternative strategies that will maximize the ability to socially distance for those who test PCR positive; 5) Supportive counseling.
  Arms: onsite Point-of-care (o-POC)

SUMMARY:
Given the likelihood of COVID-19 remaining an endemic disease among high-risk populations, establishing effective mitigation interventions will be critical to stemming community transmission. Criminal justice-involved individuals are extremely important to reducing community-based SARS-CoV-2 transmission due to their increased risk of contracting SARS-CoV-2 while incarcerated and their likelihood of living in congregate settings after incarceration. The investigators will evaluate an onsite Point-of-Care SARS-CoV-2 testing and education strategy in a corrections-focused community-based organization and its impact on improving testing uptake, mitigation behaviors(e.g. mask wearing, hand hygiene, social distancing, vaccine uptake when available), and cost-effectiveness.

DETAILED DESCRIPTION:
The United States(U.S.) has experienced higher mortality than any other nation due to COVID-19 with nearly 13.5 million cases and over 268,103 deaths. Due to the limited ability to socially distance, poor ventilation, and limited hygiene supplies, U.S. prisons and jails have observed explosive transmission of SARS-CoV-2 accounting for the 10 largest U.S. outbreaks. Because 95% of criminal justice-involved individuals reenter societyCOVID-19 transmission extends beyond those who are currently incarcerated. As justice-involved individuals reenter the community, they face high rates of homelessness, and many others live in other congregate settings such as converted hotels and halfway houses. The increased risk of SARS-CoV-2 while incarcerated coupled with the likelihood of living in congregate settings after incarceration, create conditions ripe for rapid COVID-19 transmission that will be critical to address in order to gain control of COVID-19 in the U.S. The goal of this study is to test the impact and cost-effectiveness of an intervention to mitigate SARS-CoV-2 transmission among justice-involved individuals recently released from incarceration. The investigators will conduct a randomized trial to compare the effectiveness of an onsite Point-of-Care SARS-CoV-2 testing and education intervention with community health workers (CHWs) as a central component compared to the standard of care at a community-based organization (CBO) that provides services to justice-involved individuals in New York City. The investigators will measure costs of testing, education, and navigation, and explore the cost-effectiveness of the onsite Point-of-Care intervention compared to the standard of care. The specific aims are to:1) Test the effectiveness of an onsite PoC SARS-CoV-2 intervention in a corrections-focused CBO; 2) Model the cost-effectiveness of an onsite PoC SARS-CoV-2 intervention among CJIs compared to SoC. Because testing, education, and navigation will be provided by CHWs in a culturally-sensitive environment and test results will be received in minutes (rather than days), the investigators hypothesize that O-PoC will be associated with improved testing uptake and receipt of test results, mitigation behaviors (mask wearing, hand hygiene, social distancing), and those who attend more O-PoC sessions will have better adherence to mitigation behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Fortune Society clients
* Greater than or equal to 18 years old
* Fluent in English or Spanish
* Resident of NYC
* Released from a jail or a prison system within 90 days

Exclusion Criteria:

* Inability to provide informed consent
* Inability to complete study visits over 12 months
* Does not plan to reside in the NYC area for the next year
* Terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Testing uptake | 12 months
  Testing uptake will be defined as the number and proportion of tests performed and will be determined using Program logs and healthcare record extraction. For all participants, the proportion of tests will be calculated from the total possible denominator of 5 tests (at times 0, 3, 6, 9, and 12 months). Receipt of test results will be defined as the number and proportion of test received and will be determined by self-report

SECONDARY OUTCOMES:
Mitigation measures | 12 months
  For mitigation measures, participants will be asked: Which of the following have you done in the last 14 days to keep yourself safe from coronavirus? Worn a mask or other face covering; Washed your hands with soap or used hand sanitizer; Avoided contact with people who could be high-risk; Avoided public spaces, gatherings, or crowds.For answers to which the answer is yes: The investigators will ask questions about mitigation measures on a sliding Likert scale regarding the last 14 days that will be programmed into Ethica software. Likert scales will include a legend with both numbers (1 day-14 days). The investigators will assign a score with higher adherence to mitigation measures as higher scores (from 1 to 14) and create a composite score averaging 2-week questionnaire conducted over the course of the 3 months following PoC intervention visits for each mitigation measure.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Akiyama, MD MSc, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (2):
- United States (2):
  - Fortune Society, Long Island City, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akiyama MJ, Spaulding AC, Rich JD. Flattening the Curve for Incarcerated Populations - Covid-19 in Jails and Prisons. N Engl J Med. 2020 May 28;382(22):2075-2077. doi: 10.1056/NEJMp2005687. Epub 2020 Apr 2. No abstract available. PMID 32240582
- [Background] Kinner SA, Young JT, Snow K, Southalan L, Lopez-Acuna D, Ferreira-Borges C, O'Moore E. Prisons and custodial settings are part of a comprehensive response to COVID-19. Lancet Public Health. 2020 Apr;5(4):e188-e189. doi: 10.1016/S2468-2667(20)30058-X. Epub 2020 Mar 17. No abstract available. PMID 32197116
- [Background] Lim YW, Andersen R, Leake B, Cunningham W, Gelberg L. How accessible is medical care for homeless women? Med Care. 2002 Jun;40(6):510-20. doi: 10.1097/00005650-200206000-00008. PMID 12021677
- [Background] Reinhart E, Chen DL. Incarceration And Its Disseminations: COVID-19 Pandemic Lessons From Chicago's Cook County Jail. Health Aff (Millwood). 2020 Aug;39(8):1412-1418. doi: 10.1377/hlthaff.2020.00652. Epub 2020 Jun 4. PMID 32496864
- [Background] USICH. Connecting People Returning from Incarceration with Housing and Homelessness Assistance. United States Interagency Council on Homelessness;2016.
- [Background] Levanon Seligson A, Parvez FM, Lim S, Singh T, Mavinkurve M, Harris TG, Kerker BD. Public Health and Vulnerable Populations: Morbidity and Mortality Among People Ever Incarcerated in New York City Jails, 2001 to 2005. J Correct Health Care. 2017 Oct;23(4):421-436. doi: 10.1177/1078345817727527. Epub 2017 Oct 5. PMID 28982284
- [Background] Lim S, Seligson AL, Parvez FM, Luther CW, Mavinkurve MP, Binswanger IA, Kerker BD. Risks of drug-related death, suicide, and homicide during the immediate post-release period among people released from New York City jails, 2001-2005. Am J Epidemiol. 2012 Mar 15;175(6):519-26. doi: 10.1093/aje/kwr327. Epub 2012 Feb 13. PMID 22331462
- [Background] Gu T, Mack JA, Salvatore M, Prabhu Sankar S, Valley TS, Singh K, Nallamothu BK, Kheterpal S, Lisabeth L, Fritsche LG, Mukherjee B. Characteristics Associated With Racial/Ethnic Disparities in COVID-19 Outcomes in an Academic Health Care System. JAMA Netw Open. 2020 Oct 1;3(10):e2025197. doi: 10.1001/jamanetworkopen.2020.25197. PMID 33084902
- [Background] Hawkins RB, Charles EJ, Mehaffey JH. Socio-economic status and COVID-19-related cases and fatalities. Public Health. 2020 Dec;189:129-134. doi: 10.1016/j.puhe.2020.09.016. Epub 2020 Oct 17. PMID 33227595
- [Background] Puglisi L, Calderon JP, Wang EA. What Does Health Justice Look Like for People Returning from Incarceration? AMA J Ethics. 2017 Sep 1;19(9):903-910. doi: 10.1001/journalofethics.2017.19.9.ecas4-1709. PMID 28905731
- [Background] Wang EA, White MC, Jamison R, Goldenson J, Estes M, Tulsky JP. Discharge planning and continuity of health care: findings from the San Francisco County Jail. Am J Public Health. 2008 Dec;98(12):2182-4. doi: 10.2105/AJPH.2007.119669. Epub 2008 Apr 1. PMID 18381994
- [Background] Walsh-Felz D, Westergaard R, Waclawik G, Pandhi N. "Service with open arms": enhancing community healthcare experiences for individuals with a history of incarceration. Health Justice. 2019 Dec 19;7(1):20. doi: 10.1186/s40352-019-0101-1. PMID 31858291
- [Background] Valera P, Boyas JF, Bernal C, Chiongbian VB, Chang Y, Shelton RC. A Validation of the Group-Based Medical Mistrust Scale in Formerly Incarcerated Black and Latino Men. Am J Mens Health. 2018 Jul;12(4):844-850. doi: 10.1177/1557988316645152. Epub 2016 May 4. PMID 27192716
- [Background] Kutnick AH, Leonard NR, Gwadz MV. "Like I Have No Choice": A Qualitative Exploration of HIV Diagnosis and Medical Care Experiences While Incarcerated and Their Effects. Behav Med. 2019 Apr-Jun;45(2):153-165. doi: 10.1080/08964289.2019.1591338. PMID 31343965
- [Background] Cutler DM, Summers LH. The COVID-19 Pandemic and the $16 Trillion Virus. JAMA. 2020 Oct 20;324(15):1495-1496. doi: 10.1001/jama.2020.19759. No abstract available. PMID 33044484
- [Background] Franco-Paredes C, Jankousky K, Schultz J, Bernfeld J, Cullen K, Quan NG, Kon S, Hotez P, Henao-Martinez AF, Krsak M. COVID-19 in jails and prisons: A neglected infection in a marginalized population. PLoS Negl Trop Dis. 2020 Jun 22;14(6):e0008409. doi: 10.1371/journal.pntd.0008409. eCollection 2020 Jun. No abstract available. PMID 32569274
- [Background] Saloner B, Parish K, Ward JA, DiLaura G, Dolovich S. COVID-19 Cases and Deaths in Federal and State Prisons. JAMA. 2020 Aug 11;324(6):602-603. doi: 10.1001/jama.2020.12528. PMID 32639537
- [Background] Schneider EC. Failing the Test - The Tragic Data Gap Undermining the U.S. Pandemic Response. N Engl J Med. 2020 Jul 23;383(4):299-302. doi: 10.1056/NEJMp2014836. Epub 2020 May 15. No abstract available. PMID 32412704
- [Background] Ali S, Asaria M, Stranges S. COVID-19 and inequality: are we all in this together? Can J Public Health. 2020 Jun;111(3):415-416. doi: 10.17269/s41997-020-00351-0. Epub 2020 Jun 23. No abstract available. PMID 32578185
- [Background] Mizumoto K, Kagaya K, Zarebski A, Chowell G. Estimating the asymptomatic proportion of coronavirus disease 2019 (COVID-19) cases on board the Diamond Princess cruise ship, Yokohama, Japan, 2020. Euro Surveill. 2020 Mar;25(10):2000180. doi: 10.2807/1560-7917.ES.2020.25.10.2000180. PMID 32183930
- [Background] Solomon L, Montague BT, Beckwith CG, Baillargeon J, Costa M, Dumont D, Kuo I, Kurth A, Rich JD. Survey finds that many prisons and jails have room to improve HIV testing and coordination of postrelease treatment. Health Aff (Millwood). 2014 Mar;33(3):434-42. doi: 10.1377/hlthaff.2013.1115. PMID 24590942
- [Background] Ott IM, Strine MS, Watkins AE, Boot M, Kalinich CC, Harden CA. Simply saliva: stability of SARS-CoV-2 detection negates the need for expensive collection devices. medRxiv 2020080320165233;
- [Background] Bannan CL, Lynch PA, Conroy EP, O'Dea S, Surah S, Betts-Symonds G, Lyons FE. Point-of-care testing for HIV in an Irish prison setting: results from three major Irish prisons. Int J STD AIDS. 2016 Oct;27(11):950-4. doi: 10.1177/0956462415601340. Epub 2015 Sep 16. PMID 26378194
- [Background] Beckwith CG, Atunah-Jay S, Cohen J, Macalino G, Poshkus M, Rich JD, Flanigan TP, Lally MA. Feasibility and acceptability of rapid HIV testing in jail. AIDS Patient Care STDS. 2007 Jan;21(1):41-7. doi: 10.1089/apc.2006.006. PMID 17263656
- [Background] Beckwith CG, Kurth AE, Bazerman LB, Patry EJ, Cates A, Tran L, Noska A, Kuo I. A pilot study of rapid hepatitis C virus testing in the Rhode Island Department of Corrections. J Public Health (Oxf). 2016 Mar;38(1):130-7. doi: 10.1093/pubmed/fdv023. Epub 2015 Mar 2. PMID 25736438
- [Background] Wolters F, van de Bovenkamp J, van den Bosch B, van den Brink S, Broeders M, Chung NH, Favie B, Goderski G, Kuijpers J, Overdevest I, Rahamat-Langedoen J, Wijsman L, Melchers WJ, Meijer A. Multi-center evaluation of cepheid xpert(R) xpress SARS-CoV-2 point-of-care test during the SARS-CoV-2 pandemic. J Clin Virol. 2020 Jul;128:104426. doi: 10.1016/j.jcv.2020.104426. Epub 2020 May 11. PMID 32417674
- [Background] Frank JW, Wang EA, Nunez-Smith M, Lee H, Comfort M. Discrimination based on criminal record and healthcare utilization among men recently released from prison: a descriptive study. Health Justice. 2014 Mar 25;2:6. doi: 10.1186/2194-7899-2-6. PMID 25642407
- [Background] Wang EA, Hong CS, Samuels L, Shavit S, Sanders R, Kushel M. Transitions clinic: creating a community-based model of health care for recently released California prisoners. Public Health Rep. 2010 Mar-Apr;125(2):171-7. doi: 10.1177/003335491012500205. PMID 20297743
- [Background] Fox AD, Anderson MR, Bartlett G, Valverde J, Starrels JL, Cunningham CO. Health outcomes and retention in care following release from prison for patients of an urban post-incarceration transitions clinic. J Health Care Poor Underserved. 2014 Aug;25(3):1139-52. doi: 10.1353/hpu.2014.0139. PMID 25130230
- [Background] Wang EA, Hong CS, Shavit S, Sanders R, Kessell E, Kushel MB. Engaging individuals recently released from prison into primary care: a randomized trial. Am J Public Health. 2012 Sep;102(9):e22-9. doi: 10.2105/AJPH.2012.300894. Epub 2012 Jul 19. PMID 22813476
- [Background] Collica-Cox K. Female Offenders, HIV Peer Programs, and Attachment: The Importance of Prison-Based Civilian Staff in Creating Opportunities to Cultivate Prosocial Behaviors. Int J Offender Ther Comp Criminol. 2018 Feb;62(2):524-550. doi: 10.1177/0306624X16650680. Epub 2016 May 23. PMID 27220362
- [Background] Collica-Cox K. Counting down: HIV prison-based peer education programs and their connection to reduced disciplinary infractions. Int J Offender Ther Comp Criminol. 2014 Aug;58(8):931-52. doi: 10.1177/0306624X13490660. Epub 2013 Jun 11. PMID 23757321
- [Background] Cunningham WE, Weiss RE, Nakazono T, Malek MA, Shoptaw SJ, Ettner SL, Harawa NT. Effectiveness of a Peer Navigation Intervention to Sustain Viral Suppression Among HIV-Positive Men and Transgender Women Released From Jail: The LINK LA Randomized Clinical Trial. JAMA Intern Med. 2018 Apr 1;178(4):542-553. doi: 10.1001/jamainternmed.2018.0150. PMID 29532059
- [Background] Ballard M, Bancroft E, Nesbit J, Johnson A, Holeman I, Foth J, Rogers D, Yang J, Nardella J, Olsen H, Raghavan M, Panjabi R, Alban R, Malaba S, Christiansen M, Rapp S, Schechter J, Aylward P, Rogers A, Sebisaho J, Ako C, Choudhury N, Westgate C, Mbeya J, Schwarz R, Bonds MH, Adamjee R, Bishop J, Yembrick A, Flood D, McLaughlin M, Palazuelos D. Prioritising the role of community health workers in the COVID-19 response. BMJ Glob Health. 2020 Jun;5(6):e002550. doi: 10.1136/bmjgh-2020-002550. PMID 32503889
- [Background] Bhaumik S, Moola S, Tyagi J, Nambiar D, Kakoti M. Community health workers for pandemic response: a rapid evidence synthesis. BMJ Glob Health. 2020 Jun;5(6):e002769. doi: 10.1136/bmjgh-2020-002769. PMID 32522738
- [Background] Peretz PJ, Islam N, Matiz LA. Community Health Workers and Covid-19 - Addressing Social Determinants of Health in Times of Crisis and Beyond. N Engl J Med. 2020 Nov 5;383(19):e108. doi: 10.1056/NEJMp2022641. Epub 2020 Sep 23. No abstract available. PMID 32966715
- [Background] Counihan H, Harvey SA, Sekeseke-Chinyama M, Hamainza B, Banda R, Malambo T, Masaninga F, Bell D. Community health workers use malaria rapid diagnostic tests (RDTs) safely and accurately: results of a longitudinal study in Zambia. Am J Trop Med Hyg. 2012 Jul;87(1):57-63. doi: 10.4269/ajtmh.2012.11-0800. PMID 22764292
- [Background] Boyce MR, Menya D, Turner EL, Laktabai J, Prudhomme-O'Meara W. Evaluation of malaria rapid diagnostic test (RDT) use by community health workers: a longitudinal study in western Kenya. Malar J. 2018 May 18;17(1):206. doi: 10.1186/s12936-018-2358-6. PMID 29776359
- [Background] Xiao J, Shiu EYC, Gao H, Wong JY, Fong MW, Ryu S, Cowling BJ. Nonpharmaceutical Measures for Pandemic Influenza in Nonhealthcare Settings-Personal Protective and Environmental Measures. Emerg Infect Dis. 2020 May;26(5):967-975. doi: 10.3201/eid2605.190994. Epub 2020 May 17. PMID 32027586
- [Background] Lyu W, Wehby GL. Community Use Of Face Masks And COVID-19: Evidence From A Natural Experiment Of State Mandates In The US. Health Aff (Millwood). 2020 Aug;39(8):1419-1425. doi: 10.1377/hlthaff.2020.00818. Epub 2020 Jun 16. PMID 32543923
- [Background] Greenhalgh T, Schmid MB, Czypionka T, Bassler D, Gruer L. Face masks for the public during the covid-19 crisis. BMJ. 2020 Apr 9;369:m1435. doi: 10.1136/bmj.m1435. No abstract available. PMID 32273267
- [Background] Jefferson T, Del Mar C, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Nair S, Foxlee R, Rivetti A. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD006207. doi: 10.1002/14651858.CD006207.pub3. PMID 20091588
- [Background] Matrajt L, Leung T. Evaluating the Effectiveness of Social Distancing Interventions to Delay or Flatten the Epidemic Curve of Coronavirus Disease. Emerg Infect Dis. 2020 Aug;26(8):1740-1748. doi: 10.3201/eid2608.201093. Epub 2020 Apr 28. PMID 32343222
- [Background] MacIntyre CR, Cauchemez S, Dwyer DE, Seale H, Cheung P, Browne G, Fasher M, Wood J, Gao Z, Booy R, Ferguson N. Face mask use and control of respiratory virus transmission in households. Emerg Infect Dis. 2009 Feb;15(2):233-41. doi: 10.3201/eid1502.081167. PMID 19193267
- [Background] Alsan M, Stantcheva S, Yang D, Cutler D. Disparities in Coronavirus 2019 Reported Incidence, Knowledge, and Behavior Among US Adults. JAMA Netw Open. 2020 Jun 1;3(6):e2012403. doi: 10.1001/jamanetworkopen.2020.12403. PMID 32556260
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Frimpong JA, Shiu-Yee K, Tross S, D'Aunno T, Perlman DC, Strauss SM, Schackman BR, Feaster DJ, Metsch LR. Bundling Rapid Human Immunodeficiency Virus and Hepatitis C Virus Testing to Increase Receipt of Test Results: A Randomized Trial. Med Care. 2020 May;58(5):445-452. doi: 10.1097/MLR.0000000000001311. PMID 32040038
- [Background] Frimpong JA, D'Aunno T, Perlman DC, Strauss SM, Mallow A, Hernandez D, Schackman BR, Feaster DJ, Metsch LR. On-site bundled rapid HIV/HCV testing in substance use disorder treatment programs: study protocol for a hybrid design randomized controlled trial. Trials. 2016 Mar 3;17(1):117. doi: 10.1186/s13063-016-1225-4. PMID 26936623
- [Background] Rosenberg ES, Dufort EM, Blog DS, Hall EW, Hoefer D, Backenson BP, Muse AT, Kirkwood JN, St George K, Holtgrave DR, Hutton BJ, Zucker HA; New York State Coronavirus 2019 Response Team. COVID-19 Testing, Epidemic Features, Hospital Outcomes, and Household Prevalence, New York State-March 2020. Clin Infect Dis. 2020 Nov 5;71(8):1953-1959. doi: 10.1093/cid/ciaa549. PMID 32382743
- [Background] Jing QL, Liu MJ, Zhang ZB, Fang LQ, Yuan J, Zhang AR, Dean NE, Luo L, Ma MM, Longini I, Kenah E, Lu Y, Ma Y, Jalali N, Yang ZC, Yang Y. Household secondary attack rate of COVID-19 and associated determinants in Guangzhou, China: a retrospective cohort study. Lancet Infect Dis. 2020 Oct;20(10):1141-1150. doi: 10.1016/S1473-3099(20)30471-0. Epub 2020 Jun 17. PMID 32562601
- [Background] Dinnes J, Deeks JJ, Adriano A, Berhane S, Davenport C, Dittrich S, Emperador D, Takwoingi Y, Cunningham J, Beese S, Dretzke J, Ferrante di Ruffano L, Harris IM, Price MJ, Taylor-Phillips S, Hooft L, Leeflang MM, Spijker R, Van den Bruel A; Cochrane COVID-19 Diagnostic Test Accuracy Group. Rapid, point-of-care antigen and molecular-based tests for diagnosis of SARS-CoV-2 infection. Cochrane Database Syst Rev. 2020 Aug 26;8(8):CD013705. doi: 10.1002/14651858.CD013705. PMID 32845525
- [Background] Pasomsub E, Watcharananan SP, Boonyawat K, Janchompoo P, Wongtabtim G, Suksuwan W, Sungkanuparph S, Phuphuakrat A. Saliva sample as a non-invasive specimen for the diagnosis of coronavirus disease 2019: a cross-sectional study. Clin Microbiol Infect. 2021 Feb;27(2):285.e1-285.e4. doi: 10.1016/j.cmi.2020.05.001. Epub 2020 May 15. PMID 32422408
- See also: Johns Hopkins University. COVID-19 Dashboard by the Center for Systems Science and Engineering (CSSE) at Johns Hopkins University (JHU) — https://coronavirus.jhu.edu/map.html
- See also: Federal Bureau of Prisons - Inmate Ethnicity Statistics — https://www.bop.gov/about/statistics/statistics_inmate_ethnicity.jsp
- See also: The Marshall Project. A State-by-State Look at Coronavirus in Prisons — https://www.themarshallproject.org/2020/05/01/a-state-by-state-look-at-coronavirus-in-prisons
- See also: American Civil Liberties Union. COVID-19 Model Finds Nearly 100,000 More Deaths Than Current Estimates, Due to Failures to Reduce Jails — https://www.aclu.org/sites/default/files/field_document/aclu_covid19-jail-report_2020-8_1.pdf
- See also: Prison Policy Initiative - Jails versus Prison — https://www.prisonpolicy.org/blog/2020/05/14/jails-vs-prison-update/
- See also: Covid-19: Testing Inequality in New York City — http://www.columbia.edu/~mu2166/stu_covid19/slides_stu_covid19.pdf
- See also: No COVID-19 tests available for prisoners at center of New York outbreak, court documents show — https://abcnews.go.com/Health/covid-19-tests-prisoners-center-york-outbreak-court/story?id=69969077
- See also: Audit of Brooklyn federal jail claims lack of COVID-19 tests may have masked size of outbreak New York Daily News. — https://www.nydailynews.com/new-york/ny-brooklyn-mdc-covid-19-testing-shortage-oig-report-20201110-mniz4ygxnbbglhrjotaxin4tfq-story.html
- See also: Nelson J. House Appropriations Committee Approves '21 Funding for DOJ Programs — https://csgjusticecenter.org/house-appropriations-committee-approves-21-funding-for-doj-programs/
- See also: Cepheid. Sars-cov-2-test-development-information — https://www.cepheid.com/coronavirus
- See also: Evidence-Based, Cost-Effective Interventions To Suppress The COVID-19 Pandemic: A Systematic Review — https://www.medrxiv.org/content/10.1101/2020.04.20.20054726v2.
- See also: Facemasks and similar barriers to prevent respiratory illness such as COVID-19 — https://www.medrxiv.org/content/10.1101/2020.04.01.20049528v1.
- See also: The Institute for Health Metrics and Evaluation - Daily deaths during the pandemic — https://covid19.healthdata.org/united-states-of-america?view=daily-deaths&tab=trend.
- See also: The National Reentry Resource Center. Reentry Services Directory — https://nationalreentryresourcecenter.org/reentry-services-directory/
- See also: Estimating QALY losses associated with deaths in hospital (COVID-19) — https://avalonecon.com/wp-content/uploads/2020/04/COVID-19-QALYs-v3.pdf.

DOCUMENTS (1):
  • Informed Consent Form (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT04878328/ICF_000.pdf